CLINICAL TRIAL: NCT06821165
Title: Validity and Reliability Analysis of the Dr. Goniometer Application in Elbow Flexion Measurements
Brief Title: Validity and Reliability of Dr. Goniometer in Elbow Flexion
Status: Not yet recruiting | Type: Observational
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Yasemin Şahbaz, Assistant Professor, University of Beykent
Other Study IDs: UBeykent-12
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Elbow Joint Injuries
MeSH Terms: conditions — Elbow Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elbow Flexion Measurement Group: Participants in this group will undergo elbow flexion range of motion (ROM) assessment using both a manual goniometer and the Dr. Goniometer application. Each participant's measurements will be taken twice. The measurements will be conducted twice by two different evaluators, and the average values will be analyzed to determine the validity and reliability of the Dr. Goniometer application compared to the manual goniometer.
  Interventions: Other: Dr. Goniometer Application

INTERVENTIONS:
Other: Dr. Goniometer Application — The Dr. Goniometer application is a digital tool used for measuring elbow flexion range of motion (ROM). In this study, participants' elbow flexion ROM will be assessed using both the Dr. Goniometer application and a manual goniometer. Measurements will be taken twice by two different raters to evaluate the validity and reliability of the digital application compared to the manual goniometer.

SUMMARY:
This study aims to evaluate the validity and reliability of the Dr. Goniometer application for measuring elbow flexion by comparing it with a manual goniometer. Conducted at Beykent University, the study will include 60 participants without upper extremity issues. Measurements will be taken on the dominant arm using both a manual goniometer and Dr. Goniometer, each repeated twice. Dr. Goniometer measurements will be performed twice by two different evaluators. Validity will be assessed using the Pearson correlation coefficient, while reliability will be evaluated with ICC and SEM. Measurement differences will be analyzed using a paired t-test. The results will contribute to determining the clinical applicability of the Dr. Goniometer application.

DETAILED DESCRIPTION:
This study is designed to assess both the validity and reliability of the Dr. Goniometer application for measuring elbow flexion. To do this, the study will compare the measurements taken using the Dr. Goniometer with those obtained using a manual goniometer, which is the standard tool typically used for such measurements.

Study Design and Participants:

The research will be conducted at Beykent University and will involve 60 participants. These individuals will be healthy and will not have any upper extremity issues (meaning they do not have any conditions affecting their arms).

The dominant arm of each participant will be used for measurement purposes. The dominant arm is the arm most commonly used for tasks like writing or eating.

Measurement Process:

Each participant's elbow flexion will be measured using both the manual goniometer and the Dr. Goniometer application.

The measurements will be taken twice using each tool, ensuring that there is a repetition for both the Dr. Goniometer and the manual goniometer.

Additionally, the Dr. Goniometer measurements will be performed twice by two different evaluators. This step is included to ensure that the measurements are consistent and to assess inter-rater reliability (the degree to which two different evaluators get the same results).

Statistical Analysis:

Validity will be assessed by calculating the Pearson correlation coefficient. This coefficient will measure the degree to which the measurements from the Dr. Goniometer correspond to the measurements from the manual goniometer. A high correlation would indicate that the Dr. Goniometer is valid and produces results similar to the established manual goniometer.

Reliability will be evaluated using two methods:

Intraclass Correlation Coefficient (ICC): This will assess the consistency or agreement of measurements taken with the same tool (e.g., using the Dr. Goniometer application multiple times by the same or different evaluators).

Standard Error of Measurement (SEM): This will measure the precision of the measurements and help understand the typical error expected in the measurements.

Measurement differences between the two tools (Dr. Goniometer and manual goniometer) will be analyzed using a paired t-test. This test will help determine whether there are any statistically significant differences between the measurements obtained from the two devices. If there is a significant difference, it could suggest that one tool is more accurate than the other or that they produce inconsistent results.

Expected Outcome:

The study will aim to determine whether the Dr. Goniometer application is clinically applicable. By assessing both its validity (how well it measures what it is intended to measure) and its reliability (how consistent and precise it is), the results will provide insight into whether this mobile application can be used effectively in clinical settings as a tool for measuring elbow flexion. If the application is found to be both valid and reliable, it could offer a convenient and accessible alternative to the traditional manual goniometer.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years
* No history of musculoskeletal, neurological, or orthopedic conditions
* Voluntary participation

Exclusion Criteria:

* History of musculoskeletal, neurological, or orthopedic disorders affecting the upper extremity.
* Previous upper extremity trauma, surgery, or chronic pain limiting range of motion.
* Inability to provide informed consent or follow verbal instructions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of healthy adults aged 18-65 who have no history of musculoskeletal, neurological, or orthopedic disorders affecting the upper extremity. Participants will be recruited voluntarily from the general population and must be able to provide informed consent and follow verbal instructions.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Validity and Reliability of Dr. Goniometer in Elbow Flexion Measurements | Baseline
  Comparison of elbow flexion range of motion measurements obtained using the Dr. Goniometer application and a universal goniometer to assess validity and reliability. Measurements will be taken by three independent raters, and intra-rater and inter-rater reliability will be analyzed using ICC and SEM. Pearson correlation will be used to determine validity.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gajdosik RL, Bohannon RW. Clinical measurement of range of motion. Review of goniometry emphasizing reliability and validity. Phys Ther. 1987 Dec;67(12):1867-72. doi: 10.1093/ptj/67.12.1867. PMID 3685114
- [Background] Jee H, Park J. Comparative Analyses of the Dominant and Non-Dominant Upper Limbs during the Abduction and Adduction Motions. Iran J Public Health. 2019 Oct;48(10):1768-1776. PMID 31850253
- [Background] Rothstein JM, Miller PJ, Roettger RF. Goniometric reliability in a clinical setting. Elbow and knee measurements. Phys Ther. 1983 Oct;63(10):1611-5. doi: 10.1093/ptj/63.10.1611. PMID 6622536